CLINICAL TRIAL: NCT05249972
Title: A Randomized Phase III, Three-parallel Arm, Assessor Blind, Multi-centre Study to Evaluate the Efficacy, Safety and Tolerability of AKP02 Cutaneous Spray Versus Enstilar Cutaneous Foam in Subjects With Mild to Moderate Psoriasis.
Brief Title: A Phase III Study in Subjects With Mild to Moderate Psoriasis.
Acronym: AKVANO-AKP02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lipidor AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRSC20008
Record Dates: First submitted 2022-01-29; First posted 2022-02-22 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Mild to Moderate Psoriasis
MeSH Terms: interventions — calcipotriene; Betamethasone

STUDY DESIGN:
Intervention Model Description: A randomized, assessor blind, parallel group, three arms, active and placebo controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AKP02 (Experimental): cutaneous spray (calcipotriol 50 μg/g + betamethasone 0.5 mg/g/ AKVANO)
  Interventions: Drug: AKP02/AKVANO cutaneous spray (calcipotriol 50 μg/g + betamethasone 0.5 mg/g/ AKVANO); Drug: Enstilar Topical Product (calcipotriol 50 μg/g + betamethasone 0.5 mg/g); Other: Placebo
- Enstilar (Active Comparator): cutaneous foam (calcipotriol 50 μg/g + betamethasone 0.5 mg/g)
  Interventions: Drug: AKP02/AKVANO cutaneous spray (calcipotriol 50 μg/g + betamethasone 0.5 mg/g/ AKVANO); Drug: Enstilar Topical Product (calcipotriol 50 μg/g + betamethasone 0.5 mg/g); Other: Placebo
- Placebo (Placebo Comparator): cutaneous spray
  Interventions: Drug: AKP02/AKVANO cutaneous spray (calcipotriol 50 μg/g + betamethasone 0.5 mg/g/ AKVANO); Drug: Enstilar Topical Product (calcipotriol 50 μg/g + betamethasone 0.5 mg/g); Other: Placebo

INTERVENTIONS:
Drug: AKP02/AKVANO cutaneous spray (calcipotriol 50 μg/g + betamethasone 0.5 mg/g/ AKVANO) — Topical cutaneous spray
Drug: Enstilar Topical Product (calcipotriol 50 μg/g + betamethasone 0.5 mg/g) — Topical foam
Other: Placebo — Placebo cutaneous spray

SUMMARY:
A randomized, assessor blind, parallel group, three arms, active and placebo controlled study with objective to demonstrate therapeutic non-inferiority of AKP02 cutaneous spray (calcipotriol 50 μg/g + betamethasone 0.5 mg/g/ AKVANO) versus Enstilar cutaneous foam (calcipotriol 50 μg/g + betamethasone 0.5 mg/g) in subjects with mild to moderate plaque psoriasis.

DETAILED DESCRIPTION:
Eligible subjects (in total 294) will be randomized in a 3:3:1 fashion to receive AKP02 cutaneous spray, Enstilar cutaneous foam or the AKVANO vehicle spray, respectively. The randomization will be stratified by skin type (Fitzpatrick skin type I-III and Fitzpatrick skin type IV-VI). At least 25 % of the subjects randomized in the study should belong to Fitzpatrick skin type I-III and at least 25 % to Fitzpatrick skin type IV-VI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female subjects aged >18 years having either Fitzpatrick skin type I-III or IV-VI at the time of screening.
2. A clinical diagnosis of stable (at least 6 months) psoriasis vulgaris on body, or body and scalp, involving 5 to 10% of body surface area (BSA) and PASI ≤10., that does not include the face, axilla and groin areas.
3. Mild or moderate Psoriasis on Physician Global Assessment (PGA) score (grade 2 - 3).
4. A plaque elevation of at least moderate severity (grade ≥ 3) at the target lesion site. The most severe lesion at Baseline should be identified as the target lesion.
5. Subjects must be willing to provide written informed consent.
6. Subjects must be willing and able to understand and can comply with study requirements, apply the medication as instructed and be able to complete the study.
7. Subject must be in general good health as judged by the Investigator, based on medical history and physical examination.

Exclusion Criteria:

1. Subject with history of hypersensitivity to betamethasone or calcipotriol or any component of the test or reference product or placebo.
2. Current diagnosis of unstable forms of psoriasis in the treatment area including guttate, erythrodermic, exfoliative, or pustular psoriasis.
3. Subjects with diagnosis of mild to moderate psoriasis only in the scalp area.
4. Other inflammatory skin disease in the treatment area that may confound the evaluation of the psoriasis vulgaris (e.g., atopic dermatitis, contact dermatitis, tinea corporis and seborrheic dermatitis).
5. Presence of pigmentation, extensive scarring, pigmented lesions, or sunburn in the treatment areas, which could interfere with the rating of efficacy parameters.
6. Subject with history of psoriasis unresponsive to topical treatments.
7. Subject with psoriasis lesions predominantly on palms and soles or palmo-plantar area.
8. Subjects with the diagnosis pustulosis palmo-plantaris
9. Subject in need of systemic treatment
10. Ongoing use of other psoriasis treatment including but not limited to topical or systemic corticosteroids, other topical medications (i.e. coal tar), oral or biologic medications for the treatment of psoriasis, and UV therapy.
11. Use of oral estrogen therapy, excluding oral contraceptive pills
12. Females who are pregnant, nursing, or planning a pregnancy
13. Females of childbearing potential who do not agree to utilize an adequate form of contraception.
14. Current significant medical problems that, in the discretion of the investigator, would put the subject at significant risk
15. Use of any investigational drug within 4 weeks prior to randomization, or 5 pharmacokinetic/pharmacodynamics half-lives, if known (whichever is longer)
16. Current or past history of hypercalcemia, calcium metabolism disorder, vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders.
17. Current immunosuppression
18. Use of biologic treatment for psoriasis (e.g., infliximab, adalimumab, alefacept) within six months prior to Baseline.
19. Use of: 1) chemotherapy, or 2) radiation therapy, within three months prior to Baseline.
20. Use of: 1) immunosuppressive drugs (e.g., tacrolimus, pimecrolimus), or 2) oral retinoids, within two months prior to Baseline.
21. Use of: 1) systemic steroids, 2) systemic antibiotics, 3) other systemic antipsoriatic treatment, 4) PUVA therapy, 5) UVB therapy, or 6) systemic anti-inflammatory agents, within one month prior to Baseline.
22. Use of: 1) topical anti-psoriatic drugs (e.g., salicylic acid, anthralin, coal tar, calcipotriol, tazarotene), 2) topical corticosteroids, or 3) topical retinoids, within 2 weeks prior to Baseline.
23. Use of medicated shampoos with possible effect on psoriasis
24. Subject with positive serology tests like HIV, HCV & HBsAg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-08-11 (Estimated); Study Completion 2022-08-18 (Estimated)

PRIMARY OUTCOMES:
Percentage change in Psoriasis Area and Severity Index (PASI) score | From baseline/randomization to Week 4 (Day 29±4)
  Percentage change in Psoriasis Area and Severity Index (PASI) score from baseline/randomization to the end of treatment between test product (AKP02 cutaneous spray) and comparator product (Enstilar cutaneous foam). High score is worse

SECONDARY OUTCOMES:
Percentage change in Psoriasis Scalp Severity Index (PSSI) scores | From date of randomization until Week 4 (Day 29±4) post-randomization
  Percentage change in Psoriasis Scalp Severity Index (PSSI) scores from baseline to end of treatment. High score is worse
Change in Physician's global assessment (PGA) | From date of randomization until Week 4 (Day 29±4) post-randomization
  Change in Physician's global assessment (PGA) at end of treatment compared to baseline High score is worse
Change in Scalp Physician's global assessment (ScPGA) | From date of randomization until Week 4 (Day 29±4) post-randomization
  Change in Scalp Physician's global assessment (ScPGA) at end of treatment compared to baseline High score is worse
Frequency of adverse events and serious adverse events | From date of randomization until end of study
  Frequency of adverse events and serious adverse events or any event of clinical significance

CONTACTS AND LOCATIONS:
Overall Officials: Maria Klockare, PhD, Study Director — Lipidor AB
Locations (1):
- Lotus Multispeciality Hospital, Ahmedabad, India

IPD SHARING:
Plan to Share IPD: No
A CSR will be provide to all Investigators